CLINICAL TRIAL: NCT02218138
Title: Depression and Insulin Resistance in Adolescents
Brief Title: Learning to BREATHE: A Randomized Controlled Trial to Lower Diabetes Risk in Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-4265H; R00HD069516 (NIH)
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes; Depression; Obesity
Keywords: Adolescent; Diabetes; Depression; Obesity; Stress
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression; Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Learning 2 BREATHE (Experimental): Learning 2 BREATHE, Mindfulness-based group program
  Interventions: Behavioral: Learning 2 BREATHE
- Colorado Blues (Experimental): Colorado Blues, Cognitive-behavioral depression prevention group
  Interventions: Behavioral: Colorado Blues

INTERVENTIONS:
Behavioral: Learning 2 BREATHE — Mindfulness-based group program
  Arms: Learning 2 BREATHE
Behavioral: Colorado Blues — Colorado Blues, Cognitive-behavioral depression prevention group
  Arms: Colorado Blues

SUMMARY:
Type 2 diabetes is a chronic disease that puts people at risk for major health problems like heart disease. Type 2 diabetes is the most common type of diabetes in adults. However, there has been a concerning rise in type 2 diabetes among teenagers. Diabetes develops through poor insulin sensitivity, meaning that insulin - an important chemical the body makes to keep blood sugar normal - isn't working properly. Type 2 diabetes can be prevented by improving insulin sensitivity. Stress is related to insulin sensitivity. Individuals who feel stressed have worse insulin sensitivity than individuals who do not feel stressed. In adults, decreasing stress leads to improvements in insulin sensitivity, but this hasn't been tested in teenagers. The purpose of this study is to find out if taking part in a brief group program to decrease stress will improve insulin sensitivity and lower diabetes risk in teenage girls.

DETAILED DESCRIPTION:
After a screening to determine eligibility, girls are randomly assigned to take part in one of two 6-week group programs: 1) Learning to BREATHE - a mindfulness-based program, or 2) Colorado Blues - a cognitive-behavioral program. After the group, girls return for three follow-up visits over the course of a year. The main outcomes are depressive symptoms and insulin resistance. We also are assessing stress, eating behavior, fitness, and mindfulness.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-17 years
* Female
* Overweight or obese, defined as a body mass index (BMI; kg/m2) ≥ 85th percentile for age
* Family history of type 2 diabetes or pre-diabetes in 1st degree relative (e.g., parent or sibling) or 2nd degree relative (e.g., aunt, uncle, or grandparent)
* Elevated stress/symptoms of depression as indicated by a Center for Epidemiological Studies-Depression Scale Total Score ≥ 16
* Good general health as reported by adolescent and parent/guardian
* English speaking (required for adolescent only, because the groups will be conducted in English)

Exclusion Criteria:

* Pregnancy
* Current psychiatric disorder such as major depressive disorder necessitating treatment
* Type 2 diabetes as indicated by fasting glucose > 126 mg/dL
* Use of medication affecting insulin resistance, body weight, or mood such as anti-depressants or stimulants
* Current psychotherapy or weight loss treatment

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2013-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Homeostasis model assessment of insulin resistance | 1 year
  Derived from fasting insulin and glucose

SECONDARY OUTCOMES:
Center for Epidemiological Studies-Depression Scale | 1 year
  Total sum score reflecting a continuous measure of depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Lauren B Shomaker, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shomaker LB, Pivarunas B, Annameier SK, Gulley L, Quaglia J, Brown KW, Broderick P, Bell C. One-Year Follow-Up of a Randomized Controlled Trial Piloting a Mindfulness-Based Group Intervention for Adolescent Insulin Resistance. Front Psychol. 2019 May 8;10:1040. doi: 10.3389/fpsyg.2019.01040. eCollection 2019. PMID 31133946
- [Derived] Shomaker LB, Bruggink S, Pivarunas B, Skoranski A, Foss J, Chaffin E, Dalager S, Annameier S, Quaglia J, Brown KW, Broderick P, Bell C. Pilot randomized controlled trial of a mindfulness-based group intervention in adolescent girls at risk for type 2 diabetes with depressive symptoms. Complement Ther Med. 2017 Jun;32:66-74. doi: 10.1016/j.ctim.2017.04.003. Epub 2017 Apr 15. PMID 28619307
- See also: Adolescent Wellness Lab Website — http://awl.colostate.edu/